CLINICAL TRIAL: NCT05054530
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO ASSESS THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF GMA106 IN HEALTHY, OVERWEIGHT AND OBESE ADULTS
Brief Title: Assessment of the Safety, Tolerability, and Pharmacokinetic of GMA106
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gmax Biopharm Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Organization: Gmax Biopharm LLC. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GMA106-I-101
Record Dates: First submitted 2021-09-12; First posted 2021-09-23 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Phase 1 - divided in 2 stages:
  The 1st stage: single ascending dose (SAD) The 2nd stage: multiple ascending doses (MAD)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be double-blinded. The subjects and the clinical personnel involved in the collection, monitoring, revision, or evaluation of adverse events, or personnel who could have an impact on the outcome of the study will be blinded with respect to the subject's treatment assignment (GMA106 Injection or GMA106 placebo Injection)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMA106 (Experimental): 9 different dosages will be subcutaneously injected into the abdomen.
  Interventions: Drug: GMA106 Injection
- Matching placebo (Placebo Comparator): 9 different dosages will be subcutaneously injected into the abdomen.
  Interventions: Drug: GMA106 Matching Placebo

INTERVENTIONS:
Drug: GMA106 Injection — GMA106 solution for injection. Subjects in each cohort will receive a single injection of GMA106 or matching placebo under fasting conditions and at the following target dose levels.
  Other Names: GMA106
  Arms: GMA106
Drug: GMA106 Matching Placebo — Matching Placebo for GMA106
  Other Names: Matching placebo for GMA106
  Arms: Matching placebo

SUMMARY:
This will be a single centre, Phase 1, placebo-control, randomized, double-blind, sequential single and multiple ascending dose study to assess the safety, tolerability, and PK of GMA106 in healthy, overweight or obese subjects.

DETAILED DESCRIPTION:
The objective of the study is to assess the safety, tolerability, and PK of single and multiple GMA106 SC injection. The study design is a standard design for this type of study.

This SAD study will consist of 6 cohorts (1 cohort per dose level). Within each cohort, 8 subjects will be randomized in a 3:1 ratio to receive under fasting conditions, either the study drug GMA106, or matching placebo. In each cohort, 6 subjects will be administered GMA106 and 2 subjects will receive the matching placebo, for a total of 48 subjects planned for evaluation in this study. One randomization scheme will be produced for each cohort separately.

There will be 3 cohorts in the MAD study. Dose groups in MAD are consisted of 20 mg, 40 mg and 80mg. Subjects will be dosed once a week in fasting conditions for 12 weeks. In 20 mg multiple doses group (Cohort 7), 4 subjects will be randomized in a 3:1 ratio to receive GMA106 or matching placebo throughout the course of 12 weeks. In 40 mg (Cohort 8) and 80 mg (Cohort 9) multiple doses groups, 7 subjects will be randomized in a 6:1 ratio, respectively. A total of 18 subjects planned for evaluation in the MAD study. A randomization system will be created for the MAD study.

ELIGIBILITY:
Inclusion Criteria:

SAD:

Subjects must meet all of the following criteria:

1. Male or female.
2. ≥ 18 and ≤ 60 years of age.
3. BMI > 20.0 and < 32.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
4. Non-smoker or light-smoker (≤5 cigarettes or equivalent of nicotine per day within 2 months) prior to screening. A Light smoker must agree to abstain from smoking from screening until after the last PK blood sample collection for GMA106 (Day 30±1), ≤5 cigarettes or equivalent of nicotine are permitted after that.
5. Healthy conditions are defined as:

   1. The absence of currently significant illness and surgeries, within 4 weeks prior to study drug administration.
   2. The absence of disease history, such as diseases of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and chronic condition of the urogenital, reproductive, musculoskeletal, endocrine systems, or cancer history.
6. On top of at least one contraceptive method used by his or her partner, male or female subjects must agree to use at least one contraceptive method throughout the study period, except total abstinence from heterosexual intercourse (when this is in line with the preferred and usual lifestyle of the subjects).

   1. Female subjects with childbearing potential must agree to use at least one of the following contraceptive methods throughout the study period:

      * On top of condom used by her male partner, in case of a female subject who likes to use hormonal contraceptives, the hormone must be used 4 weeks prior to study drug administration.
      * On top of condom used by her male partner, in case of a female subject who likes to use intra-uterine contraceptive device, the device must be placed at least 4 weeks prior to study drug administration.
      * On top of condom used by her male partner, in case of a female subject who likes to use diaphragm or cervical cap, the method must be started at least 21 days prior to study drug administration.

        * Contraceptive requirements for women of non-childbearing potential are defined as:
      * Postmenopausal for 1 year, not taking hormone therapy at screening, and confirmed by FSH at screening.
      * Surgically sterile women mean women who have been surgically sterilized (defined as hysterectomy, bilateral salpingectomy AND bilateral oophorectomy). Females who have only had hysterectomy (not including bilateral salpingectomy and bilateral oophorectomy) or tubal ligation or other birth control operations are NOT included.
      * Only on this premise, surgically sterile women, or post-menopausal women are the women of non-childbearing potential, and do not need to use contraception.
   2. Male subjects must agree to use at least one of the following contraceptive methods throughout the study period:

      * On top of hormonal contraceptives or intra-uterine contraceptive devices used by his female partner at least 4 weeks prior to study drug administration, the male subject must use condoms from study drug administration.
      * On top of diaphragm or cervical cap used by his female partner, the male subject must use condoms from study drug administration.
   3. Male subjects (including men who have had a vasectomy) with a pregnant partner must agree to use a condom from study drug administration.
7. Male subjects must agree not to donate sperm throughout the study period.
8. Female subjects must agree not to donate ovules throughout the study period.
9. Participants with same-sex partners as well as abstinence from penile-vaginal intercourse are eligible for the study without needing contraception when this is their usual form of sexual relations.
10. Capable and agree to give informed consent prior to any study-specific activities/procedures.
11. Subjects must agree to maintain current general diet and physical activity regimen, except for the physical activity in the 72 hours before each blood sample collection for the clinical laboratory analysis, which should not be strenuous.

MAD:

Subjects must meet all of the following criteria:

1. Male or female.
2. ≥ 18 and ≤ 60 years of age.
3. BMI ≥ 25.0 and ≤ 40.0 kg/m2.
4. Non-smoker or light-smoker (≤5 cigarettes or equivalent of nicotine per day within 2 months) prior to screening. A Light smoker must agree to abstain from smoking from screening until checking out from the clinical site on Day 4, ≤5 cigarettes or equivalent of nicotine are permitted after that.
5. Subjects who are with diagnosis of T2DM and HbA1c ≤ 8.0% at screening are allowed, but need:

   1. Taking metformin only, with stable dose at least 3 months prior to screening. OR
   2. Taking exercise and diet control (self-reported).
6. Subjects with well-controlled comorbidities, such as hypertension, dyslipidemia, fatty liver, obstructive sleep apnea, hypothyroidism, osteoarthritis, pain disorder, reflux disease and gout, at the discretion of the investigators, are allowed.
7. Have a stable body weight (< 5 kg self-reported change during the previous 8 weeks) before screening.
8. On top of at least one contraceptive method used by his or her partner, male or female subjects must agree to use at least one contraceptive method throughout the study period, except total abstinence from heterosexual intercourse (when this is in line with the preferred and usual lifestyle of the subject).

   1. Female subjects with childbearing potential must agree to use at least one of the following contraceptive methods throughout the study period:

      * On top of condom used by her male partner, in case of a female subject who likes to use hormonal contraceptives, the hormone must be used 4 weeks prior to study drug administration.
      * On top of condom used by her male partner, in case of a female subject who likes to use intra-uterine contraceptive device, the device must be placed at least 4 weeks prior to study drug administration.
      * On top of condom used by her male partner, in case of a female subject who likes to use diaphragm or cervical cap, the method must be started at least 21 days prior to study drug administration.

        * Contraceptive requirements for women of non-childbearing potential are defined as:
      * Postmenopausal for 1 year, not taking hormone therapy at screening, and confirmed by FSH at screening.
      * Surgically sterile women means women who have been surgically sterilised (defined as hysterectomy, bilateral salpingectomy AND bilateral oophorectomy). Females who have only had hysterectomy (not including bilateral salpingectomy and bilateral oophorectomy) or tubal ligation or other birth control operations are NOT included.
      * Only on this premise, surgically sterile women, or post-menopausal women are the women of non-childbearing potential, and do not need to use contraception.
   2. Male subjects must agree to use at least one of the following contraceptive methods throughout the study period:

      * On top of hormonal contraceptives or intra-uterine contraceptive devices used by his female partner at least 4 weeks prior to study drug administration, the male subject must use condoms from study drug administration.
      * On top of diaphragm or cervical cap used by his female partner, the male subject must use condoms from study drug administration.
   3. Male subjects (including men who have had a vasectomy) with a pregnant partner must agree to use a condom from study drug administration.
9. Male subjects must agree not to donate sperm throughout the study period.
10. Female subjects must agree not to donate ovules throughout the study period.
11. Participants with same-sex partners as well as abstinence from penile-vaginal intercourse are eligible for the study without needing contraception when this is their usual form of sexual relations.
12. Capable and agree to give informed consent prior to any study-specific activities/procedures.
13. Subjects must agree to maintain current general diet and physical activity regimen, with the exception of the 72 hours preceding each blood sample collection for clinical laboratory analysis, when physical activity should not be strenuous.

Exclusion Criteria:

SAD:

Subjects who meet any of the following criteria will be excluded from the study:

1. Any clinically significant (in the opinion of the Investigator) abnormality at physical examination, abnormal laboratory test results or positive test for HIV, hepatitis B, or hepatitis C found during medical screening. Abnormal laboratory values will include: liver function tests (LFTs) > 1.5x ULN
2. Clinically significant (in the opinion of the Investigator) presence of acute illness (e.g., gastrointestinal illness, gall bladder disease [cholecystectomy is allowed], chronic pancreatitis, infection such as influenza, upper respiratory tract infection) upon admission to the study site.
3. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2).
4. History of renal impairment or renal disease and/or estimated glomerular filtration rate ≤ 90 mL/min (as calculated by Cockroft and Gault formula).
5. Positive urine drug screen, or alcohol breath test at screening or at admission, positive urine cotinine test at admission.
6. Positive pregnancy test at screening or at admission.
7. Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 160 mmHg, diastolic blood pressure lower than 50 or over 95 mmHg, or heart rate less than 45 or over 100 bpm) at screening.
8. History of type 1 hypersensitivity or severe cutaneous adverse reaction to any medication, or to any excipient in the formulation, or history of significant atopy.
9. Women who intend to become pregnant or are lactating.
10. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (average weekly alcohol intake that exceeds 10 units per week, or are unwilling to stop alcohol consumption for 24 hours prior to study treatment administration until the last PK sample collection of GMA106 of the study on Day 30±1 (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
11. History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
12. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days or 5 x T1/2 whichever is longer prior to dosing, administration of a biological product in the context of a clinical research study within 90 days or 5 x T1/2 whichever is longer prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
13. Use of medications for the timeframes specified below, with the exception of hormonal contraception, medications exempted by the Investigator on a case-by- case basis because they are judged unlikely to affect the pharmacokinetic profile of the study treatment or subject safety (e.g., topical drug products without significant systemic absorption):

    1. Prescription medications within 14 prior to study treatment administration;
    2. Over-the-counter (OTC) products and natural health products (including herbal remedies homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to study treatment administration, with the exception of the occasional use of paracetamol/acetaminophen (up to 2 g daily) and ibuprofen (up to 800 mg daily);
    3. Depot injection or implant of any drug within 3 months prior to study treatment administration.
14. Live or live attenuated vaccine within 3 months prior to study drug administration and live or live attenuated vaccine planned over the course of the study.
15. COVID-19 vaccine within 14 days prior to study drug administration and within Day 30±1 after study treatment administration.
16. Have received chronic (>14 consecutive days) systemic glucocorticoid therapy (except for topical, intra-articular and inhaled preparations) within the last 12 months or have received any glucocorticoid therapy within 30 days before screening.
17. Receiving treatment or participation in an organized weight loss program that may cause significant weight gain or loss within 3 months before screening or scheduled within the study duration period.
18. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to study treatment administration.
19. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

MAD:

Subjects who meet any of the following criteria will be excluded from the study:

1. Positive test for HIV, hepatitis B, or hepatitis C found during medical screening.
2. Clinically significant abnormal laboratory test results found during medical screening. Among which, the exclusion criteria for AST, ALT and/or total bilirubin >2 x ULN, HbA1c > 8%, fasting serum glucose > 144 mg/dL (8.0 mmol/L), and/or a triglyceride level >500 mg/dL (5.65 mmol/L).
3. Any clinically significant abnormality detected during the physical examination, at the discretion of the investigators.
4. Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 160 mmHg, diastolic blood pressure lower than 50 or over 95 mmHg, or heart rate less than 45 or over 100 bpm) at screening.
5. Currently significant illness and surgeries, within 4 weeks prior to dosing.
6. History of chronic diseases, such as diseases of neurological, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, and chronic conditions of the urogenital, reproductive, musculoskeletal systems, or cancer history.
7. Had chronic or acute pancreatitis any time prior to study entry.
8. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2).
9. History of renal impairment or renal disease and/or estimated glomerular filtration rate ≤ 90 mL/min (as calculated by Cockroft and Gault formula).
10. History of ketoacidosis or hyperosmolar state/coma.
11. Any other types of diabetes except T2DM.
12. Treated with dipeptidyl peptidase 4 (DPP-4) inhibitors, glucagon like peptide-1 receptor agonists (GLP-1 RAs), glucose-dependent insulinotropic polypeptide receptor (GIPR) agonists/antagonists, insulin or any other oral glycemic-lowering agents except metformin, within 3 months before screening.
13. Positive urine drug screen or alcohol breath test at screening or at admission; positive urine cotinine test at admission.
14. Positive pregnancy test at screening or at admission.
15. History of type 1 hypersensitivity or severe cutaneous adverse reaction to any medication, or to any excipient in the formulation; history of significant atopy.
16. Women who intend to become pregnant or are lactating.
17. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening (average weekly alcohol intake that exceeds 10 units per week); do not agree to stop alcohol consumption from 24 hours prior to study drug administration until the last PK sample collection of GMA106 of the study on Day 107±3. (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
18. History of significant drug abuse within 1 year prior to screening; use soft drugs (such as marijuana) within 3 months prior to screening; use hard drugs (such as cocaine, PCP, crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
19. Participation in a clinical research study involving an investigational or marketed drug or device within 30 days or 5 x T1/2 (whichever is longer) prior to dosing; administration of a biological product in the context of a clinical research study within 90 days or 5 x T1/2 (whichever is longer) prior to dosing; concomitant participation in an investigational study involving no drug or device administration.
20. Timeframes for using medications (including over-the-counter [OTC] or prescription medicines) are specified below, with the exception of hormonal contraception, medications that are used to treat overweight/obese comorbidities (eg metformin, antihypertensives, lipid-lowering treatments, thyroid medications, pain medications, anti-gout drug etc.), and medications exempted that unlikely to affect the PK profile of the investigational drug or the safety of the subject as determined by the Investigator on a case-by-case basis (e.g., topical drug products without significant systemic absorption):

    1. Prescription medications within 14 days prior to study drug administration.
    2. OTC products (except products for pain) and natural health products (including herbal remedies homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to study drug administration.
    3. Depot injection or implant of drug within 3 months prior to study drug administration.
21. Live or live attenuated vaccine within 3 months prior to study drug administration; live or live attenuated vaccine planned throughout the study period.
22. COVID-19 vaccine within 14 days prior to study drug administration; COVID-19 vaccine planned within 30 days after the last dose of study drug administration (Day 107±3), except permitted by the Investigator on a case-by-case basis to ensure that it is appropriate for the subject to take the vaccination.
23. Have received chronic (>14 consecutive days) systemic glucocorticoid therapy (except for topical, intra-articular and inhaled preparations) within the last 12 months or have received any form of glucocorticoid therapy within 30 days before screening.
24. Receiving weight loss treatment or participating in an organized weight loss program within 3 months before screening, or schedule the weight loss treatment or program within the study period.
25. Donate plasma within 7 days prior to study drug administration; donate or lose 50 mL to 499 mL of blood (excluding volume drawn at screening) within 30 days prior to study drug administration; donate or lose more than 499 mL of blood (excluding volume drawn at screening) within 56 days prior to study drug administration.
26. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Nature, incidence and severity of treatment emergent adverse events | up to 150±5 days post injection
  Safety & Tolerability of GMA106 of Healthy subject in SAD cohort
Nature, incidence and severity of treatment emergent adverse events | up to 227±5 days post first injection
  Safety & Tolerability of GMA106 of overweight or obese subject in MAD cohort

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of GMA106 and GMA106 total antibody following single SC administration in healthy subjects. | Up to 30±1 day for GMA106 and up to 150±5 days post injection for GMA106 total antibody
  Maximum observed concentration (Cmax)
Pharmacokinetic (PK) profile of GMA106 and GMA106 total antibody following multiple SC administration in overweight or obese subjects. | Up to 107±3 day for GMA106 and up to 227±5 days post the first injection for GMA106 total antibody
  Maximum observed concentration (Cmax)
Pharmacokinetic (PK) profile of GMA106 and GMA106 total antibody following single SC administration in healthy subjects. | Up to 30±1 day for GMA106 and up to 150±5 days post injection for GMA106 total antibody
  Area under the concentration versus time curve (AUC0-t)
Pharmacokinetic (PK) profile of GMA106 and GMA106 total antibody following multiple SC administration in overweight or obese subjects. | Up to 107±3 day for GMA106 and up to 227±5 days post the first injection for GMA106 total antibody
  Area under the concentration versus time curve (AUC0-t)
Pharmacokinetic (PK) profile of GMA106 and GMA106 total antibody following single SC administration in healthy subjects. | Up to 30±1 day for GMA106 and up to 150±5 days post injection for GMA106 total antibody
  Time of Cmax
Pharmacokinetic (PK) profile of GMA106 and GMA106 total antibody following multiple SC administration in overweight or obese subjects. | Up to 107±3 day for GMA106 and up to 227±5 days post the first injection for GMA106 total antibody
  Time of Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, Prof, Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia